CLINICAL TRIAL: NCT06531083
Title: Feasibility of PRospective Surveillance and Early PhysiCal Therapy for TrIsmuS in Individuals With Head and Neck CancEr: A Single-Group Feasibility Trial (PRECISE)
Brief Title: Feasibility of Prospective Surveillance and Early Physical Therapy for Trismus
Acronym: PRECISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-24-0240
Record Dates: First submitted 2024-07-23; First posted 2024-07-31 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Cancer; Trismus
Keywords: Physical Therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Trismus

STUDY DESIGN:
Intervention Model Description: Prospective surveillance with early intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective Surveillance for Trismus and Early Physical Therapy Intervention (Experimental): Weekly monitoring of mouth opening and jaw function. Early intervention if the participant presents with 5% or greater reduction in mouth opening compared to pre-treatment measures. Early intervention will comprise: physical therapy, home exercises and use of a jaw stretching device.
  Interventions: Behavioral: Early physical therapy intervention

INTERVENTIONS:
Behavioral: Early physical therapy intervention — Physical therapy including manual therapy, home exercises for the neck and jaw, and use of a jaw stretching device.

SUMMARY:
Trismus, or restricted jaw movement, can occur in individuals with head and neck cancer (HNC) undergoing surgery or radiation therapy. There is a paucity of research examining interventions for trismus. We aim to assess the feasibility of prospective surveillance and early intervention to mitigate trismus in individuals undergoing HNC treatment.

Method: The investigators will conduct a pilot single group feasibility study involving 30 individuals with HNC who will be undergoing radiation therapy. Participants will be identified at the HNC new patient clinic. Participants will be seen weekly during radiation therapy and will receive early intervention including manual therapy and a device-based jaw exercise regimen if presenting with 5% or greater reduction in jaw opening compared to pre-treatment.

The investigators will assess recruitment and completion rates, intervention acceptability, and data collection procedures. Descriptive statistics will summarize feasibility metrics and participant demographics. Findings will inform the design of a larger multicentre trial.

DETAILED DESCRIPTION:
1. Background and rationale : Head and neck cancers (HNCs) originate in the nasal cavity, sinuses, lips, mouth, salivary glands, throat, and larynx. Individuals undergoing treatment for HNC often develop side effects such as oral mucositis xerostomia and experience difficulties with swallowing and speech. Along with these side effects, individuals with oral and oropharyngeal cancers can develop trismus, defined as restricted mouth opening (< 35mm).The beneficial effects of early physical therapy programs in mitigating the incidence of trismus have not yet been fully established, and there are no validated protocols or guidelines regarding exercise therapy. The findings of this study will be crucial in developing effective rehabilitation strategies for patients with HNC and also will contribute to the development of tailored exercise programs and rehabilitation protocols, enabling physical therapists specifically to deliver personalized care for individuals with HNC.
2. Research question and Objectives : i. To evaluate the feasibility of a prospective surveillance approach for the early detection of trismus in patients with HNC. ii. To determine the acceptability of implementing an early physical therapy intervention which includes jaw and neck exercises, manual therapy for the jaw, and the use of a jaw device for managing trismus in individuals with HNC.
3. Methodology : This feasibility two-phase study will recruit individuals with HNC, who are undergoing or have completed radiotherapy. Phase I includes two cohorts: (1) a prospective surveillance cohort of individuals undergoing radiotherapy who are at risk of developing trismus, and (2) a post-radiotherapy cohort of individuals with established trismus. In the surveillance cohort, PT will be initiated if jaw mobility declines by >5% relative to pre-treatment baseline or reaches a threshold of ≤35 mm. Participants in the post-radiotherapy cohort with established trismus (Mouth Opening (MO) ≤35 mm) will receive PT at enrolment. The intervention will include MT and therapeutic exercise. Phase II includes a qualitative assessment of the study's acceptability and delivery. The primary outcome is feasibility, including recruitment, adherence, and completion rates. Changes in MO will be explored descriptively as a secondary outcome. Participants will be identified at the HNC new patient clinic. Participants will receive early intervention including manual therapy and a device-based jaw exercise regimen if presenting with 5% or greater reduction in jaw opening compared to pre-treatment.

Phase II includes a qualitative assessment of the study's acceptability and delivery.

The primary outcome is feasibility, including recruitment, adherence, and completion rates. Changes in MO will be explored descriptively as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of oral, oropharyngeal, or nasopharyngeal cancer
* Be scheduled to undergo cancer treatment that includes radiation therapy
* Be able to read and understand English
* Be an Alberta resident.

Exclusion Criteria:

* Previous surgery for the temporomandibular joint that is not related to the HNC diagnosis.
* Local cancer recurrence or metastatic disease.
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: completion rate | 2 years
  Number of participants completing the study.

SECONDARY OUTCOMES:
Feasibility: recruitment rate | 2 years
  Number of participants entering the study by the number of participants eligible.
Feasibility: adherence rate | 6 weeks.
  Percentage of sessions completed over the 6-week intervention period.
Maximal interincisal opening | 3 months
  The distance from the incisal border of tooth #21 to the middle of incisal border of tooth #31
Trismus symptom questionnaire | 3 months
  Revised Gothenburg Trismus Questionnaire (0-100): higher scores indicate higher symptom burden
Quality of life related to Head and Neck Cancer | 3 months
  University of Washington Quality of Life scale (scored 0 to 100): higher scores indicate better functioning.
Cervical range of motion | 3 months
  Quantification of neck range of motion: higher scores reflect better function
Neck Disability | 3 months
  Neck Disability Index (0-50): higher scores reflect more disability
Intervention effect on health status | 6 weeks
  Global rating of change scale (VAS -7 to +7)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McNeely, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta/ Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on Borealis (University of Alberta)
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available following publication of the primary paper.
Access Criteria: On request from research team